CLINICAL TRIAL: NCT05533541
Title: The Prevalence and Impact of Gastrointestinal, Urinary and Sexual Dysfunction Following Abdomino-pelvic Radiotherapy for Childhood, Teenage and Young Adult Cancers
Brief Title: Pelvic Radiation Disease in Childhood Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: University College London Hospitals (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5420
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Radiation Disease
MeSH Terms: conditions — Abnormalities, Radiation-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to characterise the impact of radiotherapy on physical symptoms and quality of life in childhood and young adult cancer survivors. This is in line with current NHS strategic priorities and an unmet clinical need to optimise aftercare in this patient group. In order to provide effective treatment strategies, the scale and impact of symptom burden requires better characterisation.

A significant proportion of adult patients suffer with gastrointestinal and urinary symptoms and sexual dysfunction following radiotherapy treatment. However there is a lack of data in the paediatric and young adult population.

We will study patients who underwent abdomino-pelvic radiotherapy, who completed treatment between 2000 and 2021 and were under the age of 24 years at the time of treatment. Patients will be recruited from The Royal Marsden Hospital, Great Ormond St Hospital and University College Hospital.

Once these patients are identified we propose to prospectively assess severity of their ongoing symptoms using an electronic questionnaire, including relevant extracts from existing validated questionnaires. Treatment and patient related factors will be extracted from patient hospital records.

A further qualitative arm of the study will be completed on a sub-set of 10 patients. We will identify appropriate patients that are willing to participate in qualitative research at the time of consenting. One-to-one interviews will be conducted to gain a better insight into their symptom burden, quality of life, patient perceptions of current services and view of currently unmet needs.

This study will provide novel data on the frequency and severity of gastrointestinal and bladder related radiotherapy toxicity in young adult cancer survivors and assess impact on sexual function and quality of life. We would then propose to use this data to focus on service improvements within the regional paediatric and TYA cancer aftercare service driven by patient experience and clinical need.

DETAILED DESCRIPTION:
This study aims to characterise the impact of abdomino-pelvic radiotherapy on physical symptoms and quality of life in childhood and young adult cancer survivors. This is in line with current NHS strategic priorities and an unmet clinical need to optimise aftercare in this patient group. In order to provide effective treatment strategies, the scale and impact of symptom burden requires better characterisation. The results of this study will equip clinicians with a better understanding of young cancer survivors' experiences and facilitate more effective communication with these vulnerable young people.

BACKGROUND:

There are around 1,800 new cancer cases in children in the UK every year and over 80% of those diagnosed will survive 5 years or more. Radiotherapy is an important component of treatment for many children and teenagers with malignant disease. While this contributes to the likelihood of cure, it can also result in adverse effects. The prevalence and impact of pelvic radiation disease (PRD) in adult cancer survivors has been widely published, however there is currently a paucity of data in the paediatric population. Following radiotherapy 50-80% of adult patients report chronic gastrointestinal symptoms affecting daily activity, with an impact on quality of life. The most common long-term consequences are increased stool frequency, urgency, rectal bleeding and faecal incontinence. Other symptoms include tenesmus, mucous discharge, steatorrhoea, bloating and flatulence. Radiotherapy induces long term changes in bowel function as a result of progressive endothelial and stem cell dysfunction which in turn induces ischaemia and fibrosis. These chronic changes can progress over decades. Radiotherapy frequently disturbs physiological function in more than one part of the gastrointestinal tract resulting in a spectrum of late effects which can be difficult to diagnose; these include small intestinal bacterial overgrowth (SIBO), bile acid malabsorption (BAM), pancreatic insufficiency, fistula formation and ulceration. Radiotherapy produces dose dependent chronic bladder toxicity with 7-20% of adult patients experiencing at least grade 3 adverse events 5 years post treatment. Severe cases may require surgical intervention to prevent obstructive nephropathy and renal impairment. Less severe impairment of bladder function may still cause urinary frequency, urgency or incontinence that diminish quality of life. Over half of adults treated for pelvic malignancies develop sexual dysfunction, which can lead to depression, anxiety, relationship conflict, and loss of self-esteem. In men, erectile dysfunction after radiotherapy is an underdiagnosed and undertreated condition which can considerably affect the quality of life for men and their partners. Sexual function in women can be affected by physical changes, including vaginal narrowing, shortening and ultimately stenosis. There may also be atrophic changes to the vaginal and perineal tissues, a decrease in vaginal secretions and increased vaginal infections. Long-term follow-up studies report vaginal dryness, dyspareunia and reduced sexual enjoyment . The Cancer Survivorship Patient Reported Outcome Measures Survey highlighted the significant psychosocial impact on younger patients (aged 16-50). However, this data is based on adult-type malignancies and impact on mental health, psychosexual identity and overall quality of life in young people remains unknown.

The Royal Marsden GIANT (Gastrointestinal And Nutrition Team) are a multi-disciplinary team for adult patients providing an invaluable service for gastrointestinal symptom control following cancer treatment. They also take a holistic assessment approach to encompass other non-gastrointestinal symptoms and refer to urology, gynaecology and psychology teams where necessary. No such specialist service exists for children and adolescents. Our data will contribute to a business case to establish a dedicated service supporting young people through the late effects of cancer treatment with a focus on gastrointestinal, urinary and sexual function. By presenting the prevalence and impact of pelvic radiation disease in childhood cancer survivors our goal is to increase awareness and education in health professionals. These are sensitive topics for young patients who may not easily divulge their symptoms or their impact without some gentle questioning. Once these issues are discussed with their treating oncologist or general practitioner, patients can be referred on for specialist care. Determining the effect of these symptoms on a young person's quality of life and mental health is essential to supporting patients holistically.

METHODOLOGY:

We propose an investigator-led, non-commercial, cross-sectional, multicentre, questionnaire study investigating the prevalence and severity of defined late effects of abdomino-pelvic radiotherapy in childhood and young adult cancer.

A further qualitative arm of the study will be completed on a sub-set of 10-25 patients, depending on groups in the sampling matrix. Patients will indicate whether they are willing to participate in qualitative research at the time of consenting. One-to-one interviews will be conducted in person or by video call to gain a better insight into their symptom burden, quality of life, patient perceptions of current services and view of currently unmet needs.

All patients meeting the inclusion/exclusion criteria will be contacted regarding questionnaire participation so there will be no selection bias. The participants for the qualitative arm will be chosen from a sampling matrix once the results of the questionnaire are available.

An analysis of the Royal Marsden Hospital patient database has identified an estimate of 150 patients that would fit the inclusion criteria over the 20-year timeframe. We expect this to extrapolate to 400-500 patients in a pan London project covering all three treatment sites. We expect the age range of patients at the time of data collection to be 1-46 years.

Once these patients are identified, patient or parental consent will be obtained by post. Demographics, diagnosis and treatment data will be collected from hospital records. The severity of their ongoing symptoms will be assessed using an amalgamation of existing symptom-specific validated questionnaires. PRO-CTCAE will be used to survey gastrointestinal symptoms, urinary symptoms and sexual dysfunction. To ensure age-appropriateness of the survey, the sexual dysfunction questionnaire will only be sent to study participants over 18 years of age at time of data collection. Health professional contact will be surveyed as well as medication requirement. Health-related quality of life will be assessed with age-appropriate PEDs-QL. Participants will be given the choice to return the questionnaire by post or complete an electronic questionnaire. This will be available through the 'PROFILES' (Patient Reported Outcomes Following Initial treatment and Long-term Evaluation of Survivorship) system. PROFILES is an online questionnaire management system and data registry for the study of the physical and psychosocial impact of cancer and its treatment on patients and survivors. The online interface of PROFILES allows patients to log on and complete the questionnaires they have been invited to, using unique log on details.

Multivariate analysis will be used to identify factors associated with the development of specific complications - both treatment related factors such as radiotherapy dose, both to target volumes and organs at risk, additional surgery or chemotherapy, and patient related factors, including age, tumour type and site. Variation in symptom prevalence and severity will be explored over an extensive follow up period (1-22 years) to determine appropriate timing of aftercare interventions. This analysis will be supported by the Royal Marsden Hospital Research Data & Statistics Unit.

A further qualitative arm of the study will be completed on a sub-set of 10-25 patients. We will identify appropriate patients that are willing to participate in qualitative research at the time of consenting. One-to-one interviews will be conducted to gain a better insight into their symptom burden, quality of life, patient perceptions of current services and view of currently unmet needs. Participants will be chosen across the age groups. Interviews will be conducted at the Royal Marsden Hospital, or over the telephone or on a video platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients who;

  1. Were treated at The Royal Marsden Hospital, Great Ormond St Hospital or University College Hospital.
  2. Received radical radiotherapy to the abdomen and / or pelvis
  3. Were treated at age 24 years or below
  4. Completed treatment between 2000 - 2021.

Exclusion Criteria:

* Patients who;

  1. Received total body irradiation (TBI) or spinal radiation
  2. Have died, moved abroad or cannot be contacted.

Max Age: 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The proposed population for the study will be patients who received abdominal and/or pelvic radiotherapy and completed treatment between 2000 and 2021. They will have been under 24 years of age at the time of treatment. They will have been treated at The Royal Marsden Hospital, Great Ormond St Hospital or University College Hospital which are the three paediatric London-based Principal Treatment Centres (PTCs).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Primary End point | 2 years
  Proportion of childhood cancer survivors treated with abdominal or pelvic radiotherapy that develop gastrointestinal, urinary or sexual dysfunction.

SECONDARY OUTCOMES:
Secondary End point 1 | 2 years
  To explore the association of childhood cancer survivors with late effects by patient and treatment variables.
Secondary End point 2 | 2 years
  To describe the change in prevalence of late effects with time from end of treatment (5-year intervals).
Secondary End point 3 | 2 years
  To describe the proportion of patients referred for subspecialist review and/or intervention.
Secondary End point 4 | 2 years
  To explore patient's perception of long-term follow up care and support received

CONTACTS AND LOCATIONS:
Overall Officials: Henry C Mandeville, MBChB/MDRes, Principal Investigator — The Royal Marsden Hospital
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided